CLINICAL TRIAL: NCT03732222
Title: Analysis, Evaluation and Comparison of Spirometric Values After the Application of the Diaphragm Muscle Stretch Technique and the Cervical Level Rotation Impulse Technique of C3-C4
Brief Title: Stretching of the Diaphragm and Cervical Impulse Technique and Its Possible Spirometric Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCH CEU 208
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Respiratory Disease
Keywords: Diaphragm; Neck; Frenic Nerve
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the masking of the evaluator has been obtained, measuring the association between the response variables at baseline and the intervention group, by means of the variance analysis (ANOVA), for each response variable separately. We have verified that there are no differences between the means of the responses at the baseline level in each assigned intervention group, so that masking at the level of the evaluator has been carried out correctly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stretching the diaphragm muscle (Experimental): The interventor places his hands on the last costal cartilages and the subject makes an inspiration and keeps his hands resisted in the expiration.
  Interventions: Procedure: Stretching the diaphragm muscle
- Impulse technique in rotation of cervical level 3 and 4 (Experimental): The thumbs position the head in a double chin and then place it with neutral flexion-extension until focusing on the level of manipulation, ipsilateral lateral flexion and contralateral rotation approximately 45 degrees.
  Interventions: Procedure: Impulse technique in rotation of cervical level 3 and 4
- Combined technique of diaphragm muscle stretch and cervical ro (Experimental): combine both previous techniques.
  Interventions: Procedure: Combined technique of diaphragm muscle stretch and cervical rotation impulse technique level 3 and 4

INTERVENTIONS:
Procedure: Stretching the diaphragm muscle — Place the hands on the last costal cartilages and maintain the ascent of the ribs in the expiration.
  Arms: Stretching the diaphragm muscle
Procedure: Impulse technique in rotation of cervical level 3 and 4 — head to double chin position and then placed with neutral flexo-extension until focusing on the level of manipulation, ipsilateral lateral flexion and contralateral rotation approximately 45 degrees.
  Arms: Impulse technique in rotation of cervical level 3 and 4
Procedure: Combined technique of diaphragm muscle stretch and cervical rotation impulse technique level 3 and 4 — The same initial position, hand placement and technique guidelines will be used, cited in each of the techniques performed in the "intervention 1" group and the "intervention 2" group.
  Arms: Combined technique of diaphragm muscle stretch and cervical ro

SUMMARY:
This study investigates the effect of two different techniques, stretching of the diaphragm and cervical level impulse technique C3-C4, in the possible spirometric changes, vital capacity (CV), maximum expiratory flow (PEF) and maximum expiratory volume (FEV). in relation to the secondary variables (age, physical activity, BMI, sex). the subjects of the study were informed and clarified doubts about it and its subsequent reading and signing of informed consent. The subjects were randomly selected to determine which intervention group they would belong to (G1: intervention group of the diaphragm muscle stretch technique, G2: intervention group of the cervical rotation rotation impulse technique C3- C4, G3: Combined technique G1 and G2, G4: control group.The evaluation technique is spirometry.The intervention protocol is as follows, first the pre-intervention spirometry is performed, then the corresponding technique (according to intervention group), then the post-intervention spirometry, the intervention technique and at 5 minutes, the intervention technique is performed.

DETAILED DESCRIPTION:
The objectives of the study are the following: 1. To evaluate the changes in the values of the simple spirometry after the application of the study techniques: muscle stretching technique of the diaphragm (G1), rotation impulse technique of the cervical level of C3- C4 (G2) and combined technique of both (G3); 2. Determine the influence of these on measurable respiratory parameters by simple spirometry; 3. Compare the spirometric values obtained after applying the study techniques (G1, G2, G3) and the control group (G4: simulation of a previous technique); and 4. Analyze the different variables measured (age, gender, weight, height, sports practice and body mass index) in the effects of the applied treatment.

ELIGIBILITY:
Inclusion Criteria:

* Accept participating in the study (signature of informed consent).
* Be in an age range between 18 and 50 years.
* Do not present any exclusion criteria.

Exclusion Criteria:

* Do not meet the inclusion criteria.
* Have obstructive and / or restrictive respiratory problems.
* Perfect transient conditions that affect the respiratory tract, such as colds, sinusitis, influenza, respiratory allergies.
* To have a history of rib fractures.
* Congenital deformities.
* To have digestive problems.
* Paying hepatitis and / or hepatobiliary lesions.
* Suffer heart disease and / or arterial hypertension.
* Have abdominal problems.
* Provide surgical scar on the abdomen, thorax and / or neck.
* Patience cancer
* Press any type of pain at the time of conducting the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-18 (Actual)

PRIMARY OUTCOMES:
forced vital capacity | a week
  volume of air that we can exhale (quickly, sustainably and maximally) after a maximum expiration from the position of maximum inspiration. It is measured in liters (L).

SECONDARY OUTCOMES:
Forced expiratory volume in the first second | a week
  Maximum expiratory volume in the first second. Volume obtained in the first second of the forced vital capacity maneuver.

OTHER OUTCOMES:
Maximum expiratory flow | a week
  peak or peak expiratory flow obtained during the forced expiratory maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Rocha Ortiz, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Valencia, Moncada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kendall FP, Mac Creary EK, Provance PG. Muscles: functional tests, posture and pain. 5th ed. Madrid: Marbán; 2007 Souchard PE. RPG Principles of global postural reeducation. 1st ed. Barcelona: Paidotribo; 2005 American Thoracic Society / European Respiratory Society. ATS / ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002; 166: 518-624.
- See also: The University CEU-Cardenal Herrera is the first private university in the Valencian Community. It belongs to the Foundation San Pablo- CEU and is the leading educational organization in Spain with three Universities all over Spain — http://www.uchceu.es

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT03732222/Prot_SAP_ICF_000.pdf